CLINICAL TRIAL: NCT01462786
Title: Phase 1, Open-Label, Crossover, Safety and Pharmacokinetic Study of ATX-101 (Sodium Deoxycholate Injection) Following Subcutaneous Injections in the Submental and Abdominal Areas
Brief Title: To Evaluate the Safety, Tolerability and to Compare the Pharmacokinetic Profile of ATX-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATX-101-11-30
Record Dates: First submitted 2011-10-17; First posted 2011-10-31 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATX-101 in abdomen area (Experimental): Crossover study in which subjects will receive 2 mg/cm2 ATX-101 in one dosing session in either the submental area or the abdomen crossing over to the alternate area for the second dosing session
  Interventions: Drug: ATX-101
- ATX-101 in submental area (Experimental): Crossover study in which subjects will receive 2 mg/cm2 ATX-101 in one dosing session in either the submental area or the abdomen crossing over to the alternate area for the second dosing session
  Interventions: Drug: ATX-101

INTERVENTIONS:
Drug: ATX-101 — 2 mg/cm2 ATX-101

SUMMARY:
The objectives of this trial are to evaluate the safety and tolerability of ATX-101 injections and to compare the pharmacokinetic profile of ATX-101 administered into subcutaneous fat in the submental area and abdomen.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of submental fat graded by the investigator as 3 or 4 using the SMF Rating Scale (Appendix C) as a guideline.
2. Sufficient submental and abdominal fat such that the protocol-specified number of injections can be safely administered.
3. Males or nonpregnant, nonlactating females who are aged 18 to 65 years, inclusive, on the date of dosing with ATX-101. Females must have a negative serum human chorionic gonadotropin (HCG) test result from a sample obtained during the screening period and after admission to the research facility for the first confinement period, but before the dose of study material. Females of postmenopausal status must not have had menses for at least one year and if younger than 55 years of age must have a serum FSH level ≥ 35 mIU/mL. Females of childbearing potential must agree to practice adequate contraception, in the judgment of the investigator, during the course of the trial.
4. A normal result on coagulation tests (PT, PTT) obtained within 28 days before subject's first dosing session.
5. Serum hemoglobin test result of 12.0 g/dL or greater and negative hepatitis B, hepatitis C, and HIV test result within 28 days before the dose of study material.
6. Ability to comply with and understand the visit schedule and all of the protocol-specified tests and procedures.
7. Medically able to undergo the administration of study material as determined by clinical and laboratory evaluations obtained within 28 days before dosing with study material for which the investigator identifies no clinically significant abnormality.
8. Signed informed consent obtained before any study-specific procedure is conducted.

Exclusion Criteria:

1. History of any intervention to treat submental or abdominal fat (e.g., liposuction, surgery, or lipolytic agents).
2. History of trauma associated with the chin, neck, or abdominal areas, which in the judgment of the investigator may affect evaluation of safety or efficacy of treatment.
3. Loose skin in the neck or chin area for which reduction in submental fat may, in the judgment of the investigator, result in a cosmetically unacceptable outcome.
4. Prominent platysmal bands at rest that interfere with the evaluation of submental fat.
5. Evidence of any cause of enlargement in the submental or abdominal area other than localized subcutaneous fat.
6. Obesity as defined by a body mass index (BMI) > 34 at the screening visit. Refer to Appendix B.
7. Any blood donation or significant blood loss within 56 days before the dose of study material or plasma donation within 7 days before the dose of study material.
8. Any medical condition (e.g., respiratory, cardiovascular, hepatic, neurological disease, uncontrolled hypertension, thyroid dysfunction), that would interfere with the assessment of safety in this trial or would compromise the ability of the subject to undergo study procedures or to give informed consent.
9. Treatment with fish oil, aspirin, or nonsteroidal anti-inflammatory agents (NSAIDS), except acetaminophen, within seven days before dosing, or any anticipated need for agents with anticoagulative effects (e.g., warfarin, heparin) during the course of the trial.
10. Treatment with oral anticoagulants (e.g., warfarin) within 30 days before dosing with study material.
11. Expected to require treatment with any systemic medication during the study period (excluding any protocol-specified treatments)
12. Treatment with radio frequency, laser procedures, chemical peels, or dermal fillers in the neck or chin area within 12 months before the first treatment session, or botulinum toxin injections in the neck or chin area within 6 months before the first treatment session.
13. History of sensitivity to any components of the study material or to topical anesthetics (e.g., lidocaine, benzocaine, novocaine).
14. History of drug or alcohol abuse, in the judgment of the investigator, within two years before the dose of study material.
15. Presence of a positive urine drug or alcohol screening test result obtained from a sample obtained during the screening period and/or after admission to the research facility for the confinement period, but before the dose of study material.
16. Previous enrollment into a trial of ATX-101.
17. Treatment with an investigational agent within 30 days before dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety of ATX-101 injections as assessed by incidence, severity and duration of AEs of ATX-101 administered into subcutaneous fat in the submental and abdomen area | 2 weeks
  This is a single center, open-label, crossover study in which subjects will receive 2 mg/cm2 ATX-101 as indicated below in one dosing session in either the submental area or the abdomen crossing over to the alternate area for the second dosing session. For the first dosing session dosing will occur on Day 0 with the 2nd dosing session occurring on Day 8. A final follow-up visit will occur on Day 14.

SECONDARY OUTCOMES:
To compare the pharmacokinetic profile (Cmax, tmax, AUC, half-life) of ATX-101 administered into subcutaneous fat in the submental and abdomen area | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD, PhD, Study Director — Kythera Biopharmaceuticals
Locations (1):
- Cetero Research, Fargo, North Dakota, United States